CLINICAL TRIAL: NCT07247825
Title: Efficacy of Therapeutic Percutaneous Electrolysis vs Laser Therapy in Supraspinatus Tendinopathy. Randomized Clinical Trial.
Brief Title: Efficacy of Therapeutic Percutaneous Electrolysis vs Laser Therapy in Supraspinatus Tendinopathy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia de Salamanca (Other)
Responsible Party: Principal Investigator, Jorge Velazquez, Principal Investigator, Universidad Pontificia de Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161125
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Tendinopathy
Keywords: electrolysis; Quality of life; pain; laser; range of motion
MeSH Terms: conditions — Tendinopathy; Pain | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Active Comparator): Laser treatment on tendinophaty shoulder.
  Interventions: Device: Laser
- Electrolysis percutaneus (Experimental): Electrolysis treatment on tendinophaty shoulder.
  Interventions: Device: Electrolysis percutaneus

INTERVENTIONS:
Device: Electrolysis percutaneus — Electrolysis percutaneus on supraspinatus tendon.
  Arms: Electrolysis percutaneus
Device: Laser — laser on supraspinatus tendon.
  Arms: Laser treatment

SUMMARY:
Supraspinatus tendinopathy (SE) is one of the main pathologies that cause functional alterations in the glenohumeral joint. It reduces the quality of life of the population suffering from this injury. This pathology is the most frequent cause of pain in this joint. Symptoms are aggravated by repetitive work performed at or above shoulder height and sports that involve movements above the head.

Single-blind randomised clinical trial. The participants in this study will be patients selected from the ValleSur physiotherapy clinic in Ávila from January to May 2026. These patients will be diagnosed beforehand by an orthopaedic surgeon through a complete series of orthopaedic and complementary diagnostic tests. Following the clinical examination conducted by the principal investigator to verify the presence of tendinopathy in the supraspinatus and identify the selection criteria in the selected participants. Ultrasound imaging will be used to select the area to be treated. A single-blind clinical trial with a randomised design will be conducted, in which the evaluator will be blinded to assess the short- and medium-term efficacy of treatment with ultrasound-guided electrolysis. The results will then be compared with another intervention already performed with laser therapy for the same pathology and at the same centre. - Common part of the treatment: Participants included in the study receive one intervention, with four evaluations: pre-intervention, post-intervention, 24 hours and one week after the intervention.

- Invasive procedure: The patient is placed in a prone position with their feet outside the treatment table. Before beginning the intervention, the physiotherapist uses sterile gloves and examines the area to be treated using a linear probe ultrasound scanner, 2D study, in B mode and Doppler, to identify the target tissue safely and guaranteein B-mode and Doppler mode, to identify the target tissue safely and ensure the effectiveness of the technique. (10) Once the target area has been located, an ultrasound palpation is performed to correlate the ultrasound image with the patient's clinical condition. This image is frozen in order to measure the distance from the skin to the target tissue and select the needle, in this case 0.30 x 25 mm in length (Agupunt, Madrid, Spain) CE. (16,17) The physiotherapist then thoroughly cleans the area using sterile gauze and 2% aqueous chlorhexidine. The ultrasound probe is placed back on the target tissue, the needle inserted into the handpiece is introduced, and the contact electrode is placed in the upper area close to the needle to close the circuit. Once positioned in the area to be treated, the CE-certified electrolysis device for the percutaneous application of EPTE® galvanic current (IONCLINICS & DEIONIC SL, Av.

Antonio Almela 29, 46250 Alcudia, Valencia, Spain), the intensity is programmed, which in this case is 360 µA, and the treatment time, 1 minute and 20 seconds, and the 'ON' button to start the technique, and the current begins to rise progressively until it reaches 360 µA. Once the intensity is reached, the time countdown begins (1 minute and 20 seconds).

ELIGIBILITY:
Inclusion Criteria:

* Signing of informed consent both to participate in the study and to undergo invasive physiotherapy techniques.
* Presence of symptoms (inflammation or pain) ≥ 4 weeks.
* Positive palpation test of the supraspinatus tendon.
* Men and women over 18 years of age.
* Score of 3 or higher on the shoulder pain analogue scale.
* Adequate cognitive ability for understanding.
* Limited range of motion.
* Rotator cuff tendinopathy confirmed by ultrasound at the study centre, either due to tendon inflammation, presence of hypoechoic areas, calcification, fibrillar disorganisation and/or neovascularisation in the supraspinatus muscle.
* Pain in the proximal lateral part of the arm that worsens with abduction.

Exclusion Criteria:

* Any related acute or chronic musculoskeletal disease that may affect the results of the study.
* Presence of neuropathic pain such as lumbar radiculopathy, which may affect the results of the study.
* Not receiving the treatment sessions and assessments of the study.
* History of glenohumeral fracture and rheumatoid arthritis.
* Rheumatic, neurological or structural polymyalgia affecting the joint.
* Pregnancy.
* Patients with cardiovascular disease.
* Patients with neurological disease.
* Local infection.
* Tumours.
* Belonephobia.
* Taking anticoagulants or antiplatelet agents.
* Infiltrative and/or rehabilitative treatment in the two months prior to recruitment.
* Treatment with another intervention during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | 1 week
  measured using the VAS scale, where 0 is the least possible pain and 10 is the greatest possible pain

SECONDARY OUTCOMES:
Range of motion | 1 week
  Shoulder mobility in the joint ranges of flexion, extension, abduction, adduction, and external and internal rotation. Measurement in degrees using a goniometer
Patient quality of life | 1 week
  DASH questionnaire The score ranges from 0, which is equivalent to having no disability, to a maximum of 100, which is equivalent to having a very severe functional limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Redondo-Alonso L, Chamorro-Moriana G, Jimenez-Rejano JJ, Lopez-Tarrida P, Ridao-Fernandez C. Relationship between chronic pathologies of the supraspinatus tendon and the long head of the biceps tendon: systematic review. BMC Musculoskelet Disord. 2014 Nov 18;15:377. doi: 10.1186/1471-2474-15-377. PMID 25408141
- [Result] Haik MN, Alburquerque-Sendin F, Moreira RF, Pires ED, Camargo PR. Effectiveness of physical therapy treatment of clearly defined subacromial pain: a systematic review of randomised controlled trials. Br J Sports Med. 2016 Sep;50(18):1124-34. doi: 10.1136/bjsports-2015-095771. Epub 2016 Jun 10. PMID 27288517
- [Result] Romero-Morales C, Bravo-Aguilar M, Abuin-Porras V, Almazan-Polo J, Calvo-Lobo C, Martinez-Jimenez EM, Lopez-Lopez D, Navarro-Flores E. Current advances and novel research on minimal invasive techniques for musculoskeletal disorders. Dis Mon. 2021 Oct;67(10):101210. doi: 10.1016/j.disamonth.2021.101210. Epub 2021 Jun 4. PMID 34099238
- [Result] Asensio-Olea L, Leiros-Rodriguez R, Marques-Sanchez MP, de Carvalho FO, Maciel LYS. Efficacy of percutaneous electrolysis for the treatment of tendinopathies: A systematic review and meta-analysis. Clin Rehabil. 2023 Jun;37(6):747-759. doi: 10.1177/02692155221144272. Epub 2022 Dec 30. PMID 36583575
- [Result] Sanchez-Sanchez JL, Calderon-Diez L, Herrero-Turrion J, Mendez-Sanchez R, Arias-Buria JL, Fernandez-de-Las-Penas C. Changes in Gene Expression Associated with Collagen Regeneration and Remodeling of Extracellular Matrix after Percutaneous Electrolysis on Collagenase-Induced Achilles Tendinopathy in an Experimental Animal Model: A Pilot Study. J Clin Med. 2020 Oct 15;9(10):3316. doi: 10.3390/jcm9103316. PMID 33076550